CLINICAL TRIAL: NCT06291051
Title: Evaluation of the Safety of Electrical Spinal Cord Stimulation in Parkinson's Patients Presenting With Painful Camptocormia
Acronym: CAMPTOSTIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/0382/HP
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electrical spinal cord stimulation in Parkinson's patients presenting with painful camptocormia (Experimental)
  Interventions: Device: Electrical spinal cord stimulation

INTERVENTIONS:
Device: Electrical spinal cord stimulation — electrical spinal cord stimulation in Parkinson's patients presenting with painful camptocormia

SUMMARY:
Camptocormia is defined by abnormal flexion of the trunk, not fixed, present when standing and walking, resolves when lying down and often complicated by lower back pain. It can be observed in numerous neurological pathologies with a prevalence ranging between 5 and 19% in Parkinson's disease. The physiopathology of camptocormia associated with PD is not completely elucidated, however several mechanisms are discussed, including muscular hypertonia, abdominal muscle dystonia, proprioceptive deficit, iatrogenics linked to dopamine agonists, and focal myopathy. Although its impact is major and greater than the main symptoms of the disease, no specific treatment has been the subject of a marketing authorization request in this indication. Its management remains difficult and usually consists of: adjusting the antiparkinsonian treatment, reducing or even eliminating dopamine agonists, resorting to botulinum toxin injections and rehabilitation, sometimes with the use of a corset. However, the results observed are most often disappointing. The benefit of more invasive techniques, such as deep brain stimulation, classically proposed in advanced forms at the stage of motor complications of PD, is discussed by certain authors. Numerous studies thus suggest that bilateral stimulation of the NST could have a significant but moderate beneficial effect on postural disorders associated with PD, in particular on camptocormia. Likewise, the results of a retrospective study recently conducted in 36 Parkinson's patients discuss the effectiveness of bi-pallidal stimulation. Furthermore, surgical interventions by arthrodesis remain invasive and cause more frequent complications in Parkinson's patients with camptocormia compared to patients with isolated degenerative spinal pathology.

Electrical spinal cord stimulation (ESS) is a validated technique in the management of chronic neuropathic pain. Several publications suggest that it could be effective on postural disorders in PD. Thus, authors report the case of a Parkinson's patient afflicted with painful camptocormia refractory to drug treatments and deep brain stimulation who benefited from EMS with a remarkable effect on pain, walking and posture. This observation is corroborated by data collected in 3 Parkinson's patients with camptocormia subjected to EMS with a beneficial effect on painful and motor symptoms. The mechanism of action could be linked to the correction of the proprioceptive deficit via ascending stimulation of the basal ganglia. On the other hand, the effectiveness of repetitive spinal cord magnetic stimulation was evaluated in a study carried out in 37 patients with camptocormia associated with PD.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease validated according to UKPDSBB clinical criteria
* Camptocormia defined by a total camptocormia angle (ACT) > 30° or a greater camptocormia angle (ACS) > 45°
* Camptocormia established for less than 2 years or recently worsening for less than 1 year.
* Persistent camptocormia despite optimal drug treatment at the time of inclusion
* Pain associated with abnormal posture: VAS ≥ 4/10 during the last 3 months
* Stable antiparkinsonian treatment for 4 weeks
* Treatment with co-analgesics stable for 4 weeks
* Criteria relating to regulation:

  * Major person
  * Affiliation to a social security scheme
  * Adult who has read and understood the information letter and signed the consent form
  * Women:

    * Of childbearing age (defined by the CTFG as a fertile woman, after menarche and until menopause, except in cases of permanent sterility (including hysterectomy, bilateral salpingectomy or bilateral oophorectomy)):
* using effective contraception according to the WHO (combined hormonal contraception (containing estrogens and progestins), progestin-only contraception, intrauterine device IUD), male or female condoms) for 1 month before inclusion and during the study And,
* presenting a negative urine pregnancy test at inclusion - Menopause: menopause according to the CTFG is defined as the absence of periods for 12 months without any other medical cause before the inclusion visit. An elevated follicle-stimulating hormone (FSH) level in the postmenopausal interval can be used to confirm a postmenopausal state in women who are not using hormonal contraception or hormone replacement therapy. However, in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.

Exclusion Criteria:

* Atypical parkinsonian syndrome
* Contraindication to surgery and anesthetic products
* Uncontrolled diabetes
* Systemic or local infection
* Major cognitive disorders: MOCA < 25
* Severe psychosis associated with Parkinson's disease
* Severe depressive syndrome: MADRS > 35
* Patient with deep brain stimulation
* Patient with a cardiac pacemaker
* Patient currently being treated by diathermy or to be treated by diathermy
* Severe substance use disorders (alcohol, drugs, medication)
* Contraindication to MRI
* Obstacle to the placement of a dorsal epidural electrode
* Dorsal myelopathy
* Severe associated scoliosis
* Severe camptocormia defined by an ACT > 80°
* Severe alteration of somesthetic evoked potentials (ESP) in the lower limbs
* Pregnant or parturient or breastfeeding woman or proven absence of contraception
* Person deprived of liberty by an administrative or judicial decision or person placed under judicial protection/under guardianship or curatorship
* History of illness or psychological or sensory abnormality likely to prevent the subject from fully understanding the conditions required for participation in the protocol or preventing them from giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the safety of electrical spinal cord stimulation in Parkinson's patients with painful camptocormia | 11 months post-operative operative
  The presence of intraoperative or postoperative adverse events, including in particular short-term postoperative complications but also any adverse event observed until the end of study visit (V7) at 10 - 11 months post-operative operative approximately.

IPD SHARING:
Plan to Share IPD: No